CLINICAL TRIAL: NCT03926403
Title: Evaluation of the Effectiveness of Hypnosis Support on Patient Perception of Outpatient Surgery Under Local Anaesthesia in the Maxillo-Facial Surgery Department of the CHU Amiens-Picardie.
Brief Title: Evaluation of the Effectiveness of Hypnosis Support on Patient Perception of Outpatient Surgery Under Local Anaesthesia
Acronym: HYPNOFACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2019_843_0007
Record Dates: First submitted 2019-04-16; First posted 2019-04-24 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Hypnosis; Local Anaesthesia; Outpatient Surgery; FACE
Keywords: hypnosis; local anaesthesia; outpatient surgery; face surgery
MeSH Terms: interventions — Anesthesia, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis (Experimental): Patients requiring facial surgery under local anaesthesia in an ultra-short circuit will benefit from experimental management based on hypnosis techniques.
  Interventions: Other: State-Trait Anxiety Inventory ("Spielberger Self-Assessment Questionnaire"); Procedure: hypnosis techniques
- conventional management (Active Comparator): Patients requiring facial surgery under local anaesthesia in an ultra-short circuit will benefit from conventional management (local anaesthesia).
  Interventions: Other: State-Trait Anxiety Inventory ("Spielberger Self-Assessment Questionnaire"); Procedure: local anaesthesia

INTERVENTIONS:
Other: State-Trait Anxiety Inventory ("Spielberger Self-Assessment Questionnaire") — Patients will be given, a State-Trait Anxiety Inventory ("Spielberger Self-Assessment Questionnaire") that will be collected on the same day. Each patient's initial anxiety score will be calculated so as to select only patients who are at least lightly anxious about their management (score ≥ 36).
Procedure: hypnosis techniques — Patients requiring facial surgery under local anaesthesia in an ultra-short circuit will benefit from experimental management based on hypnosis techniques.
  Arms: Hypnosis
Procedure: local anaesthesia — Patients requiring facial surgery under local anaesthesia in an ultra-short circuit will benefit from conventional management (local anaesthesia).
  Arms: conventional management

SUMMARY:
Many clinical trials assessing the effectiveness of hypnosis have been conducted in recent years, some of which show that hypnosis reduces pain perception better than drug treatments administered to control groups, and that it is at least as effective as other complementary therapies (such as massage, acupuncture, yoga). However, their conclusions are limited by a significant risk of bias, and further studies with rigorous methodology remain necessary. The hypothesis of this study is that hypnosis support methods can reduce anxiety in patients requiring facial surgery under local anaesthesia, and thus improve their medical management.

The purpose of this study is to evaluate the effectiveness of hypnosis support on the patient's state of anxiety before and after outpatient surgery under local anaesthesia in the Maxillofacial Surgery Department.

DETAILED DESCRIPTION:
Interventions performed under local anaesthesia may be a particular source of anxiety for some patients, and the management of surgical pain is still a real challenge. In order to avoid the side effects of medications, a lot of caregivers are turning to complementary medicines. Hypnosis in particular has long been used in the non-pharmacological management of pain and anxiety.

Many clinical trials assessing the effectiveness of hypnosis have been conducted in recent years, some of which show that hypnosis reduces pain perception better than drug treatments administered to control groups, and that it is at least as effective as other complementary therapies (such as massage, acupuncture, yoga). However, their conclusions are limited by a significant risk of bias, and further studies with rigorous methodology remain necessary. The hypothesis of this study is that hypnosis support methods can reduce anxiety in patients requiring facial surgery under local anaesthesia, and thus improve their medical management.

Patients requiring facial surgery under local anaesthesia in an ultra-short circuit will be informed of the study in consultation by the maxillofacial surgeon. If they give their informed consent, a State-Trait Anxiety Inventory ("Spielberger Self-Assessment Questionnaire") will be given to them and collected on the same day. Each patient's anxiety score will be calculated so as to select only patients who are at least lightly anxious about their management (score ≥ 36). The latter will be randomized into 2 groups, one benefiting from experimental management based on hypnosis techniques and the other benefiting from conventional management.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated under local anaesthesia in the Maxillo Facial Surgery department with ultra-short circuit
* Patient undergoing face surgery
* Patient who has received appropriate information and has provided informed consent
* Adult patient ≥ 18 years old
* Patient with a score of ≥ 36 on the initial anxiety self-assessment questionnaire

Exclusion Criteria:

* Patient under general anaesthesia
* Patients treated in conventional inpatient care or in the traditional ambulatory circuit
* Patient under guardianship or trusteeship
* Minor patient < 18 years of age
* Patient who has not provided informed consent or who cannot submit to the study protocol
* Patient suffering from cognitive disorders (ex: Alzheimer's disease)
* Patients who are deaf or hearing-impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-01-28 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
variation in Spielberger's anxiety self-assessment questionnaire score between the patient's arrival in the operating room and his departure | on the day of surgery under local anaesthesia.
  The State-Trait Anxiety Inventory (STAI) (or Spielbergers's anxiety self-assessment questionnaire) is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. The STAI measures two types of anxiety - state anxiety, or anxiety about an event, and trait anxiety, or anxiety level as a personal characteristic. Higher scores are positively correlated with higher levels of anxiety.

SECONDARY OUTCOMES:
Value reported by the patient on the Visual Analogue Pain Scale after surgery | on the day of surgery under local anaesthesia.
  The visual analogue scale (VAS) is commonly used as the outcome measure. It is usually presented as a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable."
Variation of amount of local anaesthetic | on the day of surgery under local anaesthesia.
  Amount of local anaesthetic consumed for a defined surgical procedure
measure of operating time | on the day of surgery under local anaesthesia.
  operating time for a defined surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Devauchelle, Pr, Principal Investigator — CHU Amiens; Stéphanie Dakpe, MD, Principal Investigator — CHU Amiens; Sylvie Testelin, Pr, Principal Investigator — CHU Amiens; Jérémie Bettoni, MD, Principal Investigator — CHU Amiens; Stéphanie Mauquit, N, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No